CLINICAL TRIAL: NCT02572856
Title: Continuous Glucose Monitoring During and After Surgery
Acronym: CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, David Flum, Professor, School of Medicine: Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00003457; IIS-2014-028 (Other Grant/Funding Number: Dexcom Inc)
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes
Keywords: Feasibility; continuous glucose monitor; surgery
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM patients (Experimental): Apply continuous glucose monitor, calibrate and make glucose measurements. Measurements are blinded to the care provider
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Apply Dexcom Gen 6 Professional CGM sensor at least 2.5 hours prior to surgery Configure CGM so that its measurements are blinded. Setup CGM to make continuous glucose measurements during and after surgery. Download CGM measurement data after study and compare measurements against glucose measurements made for clinical care.

SUMMARY:
During surgery and after surgery elevated blood glucose levels can lead to poor outcome such as wound infections. Current technology does not allow close monitoring of glucose levels often resulting in poor management of glucose levels. In this study, the investigators will evaluate the feasibility of using a continuous glucose monitor (Dexcom Gen 6 Professional) during and after surgery. Such a monitor has the potential of monitoring glucose levels continuously and in real-time, thus allowing better glucose management

DETAILED DESCRIPTION:
During surgery high blood glucose levels, termed hyperglycemia, are commonly encountered due to the physiological stress. Hyperglycemia has been associated with complications such as surgical site infections, adverse cardiovascular and pulmonary events. Optimal glucose control targeted at preventing hyperglycemia has been shown to reduce the risk of complications. However, performing optimal glycemic management during and after surgery is a significant challenge because varying effects of surgical stress and anesthesia interventions produce rapid changes in glucose levels. The current method of manually measuring blood glucose every hour or less is grossly inadequate to track changes in glucose levels. Continuous Glucose Monitors (CGMs) have the ability to automatically measure blood glucose levels in near continuous fashion. Integrating CGMs as part of a glycemic control protocol can lead to better management of glucose levels with fewer hyperglycemia episodes and lower glucose level variability resulting in better post-surgical outcome. The viability of using a CGM in during and after surgery has only been minimally studied, that too with older generation systems. The investigators propose a study that aims to evaluate viability of using a current generation CGM in surgery patients.

The primary goal of this study is to evaluate the feasibility and accuracy of a Continuous Glucose Monitor (CGM) in measuring blood glucose levels and trends in surgery patients. The secondary goal is to observe and analyze trends in perioperative blood glucose levels to understand the dynamic effects of surgical stress and anesthetic agents on blood glucose levels. This information will allow development of better intraoperative glucose management strategies and protocols. The specific aims of the study are outlined below:

1. Compare glucose measurements made by a next generation, investigational Continuous Glucose Monitor (Dexcom Gen 6 Professional CGM) against point of care (POC) glucose meter (Accu Chek Inform II, Roche Diagnostics), during the intraoperative and postoperative periods.
2. Correlate the trends in glucose levels measured by a CGM against surgery and anesthesia events (Induction, Incision, Emergence) and factors, and administration of anesthetic drugs (inhalational agents, steroids, etc)

The study protocol is described below:

CGM:

Dexcom Gen 6 Professional CGM will be used for the proposed study. The Gen 6 CGM is FDA approved for non-hospital use. Its use for the study will be off-label as it will be used in a hospital setting. However, for this study the CGM will be used as a secondary monitor not intended for patient care. The anesthesia provider and nurse practitioner will continue to use the existing manual glucose measurements (Point of care glucose meters or laboratory measurements) for clinical care. The measurements made by the Dexcom Gen 6 CGM will be blinded (not displayed) so that the providers and the patients cannot see or use the measured values.

The sensor will be placed on the upper arm. Sensor location will be consistent across all patients. Because CGM makes interstitial glucose measurement, any interference from IV infusions is anticipated to be minimal. However, to minimize any potential interaction with an infusion (Dextrose) the placement of the sensor will be on the arm different from the IV arm, if possible. After placement, the CGM sensor requires a warm-up period of 2 hours before which measurements cannot be made.

Study protocol:

The study will be conducted in a single phase at the University of Washington Medical Center. However, after the first 4 patients, a safety evaluation will be performed. Study will be continued only if the CGM is determined to be safe and able to make glucose measurements that are comparable to those made by the standard point of care (POC) glucose meter.

Screening and Consenting:

Potential patients will be identified through a surgery schedule report or at surgeon's clinic with assistance from PCC (Patient care coordinator) who will notify a research coordinator. The research coordinator will screen the patient to make sure that he/she meets the eligibility criteria. If a patient meets eligibility criteria, the research coordinator will approach the candidate patient either via mail or during the History & Physical visit to communicate study details and provide the consent form. If an eligible patient expresses interest, research coordinator will arrange an appointment to place the CGM sensor about 2-4 hours prior to surgery.

The research coordinator will contact (by phone/email) the patient prior to surgery to answer any study related questions and to enquire about the patient's decision to participate in the study. If the candidate patient wishes to participate, the coordinator will make arrangements to obtain signed consent and enroll the patient in the study prior to surgery.

The research coordinator will meet with the eligible patient at the time of the sensor placement and collect the signed consent form, thus officially enrolling the patient for the study. The patient will be given a gift card ($50) as a token of appreciation for enrolling in the study.

Placement of the CGM sensor and calibration:

The CGM sensor has a warm-up period of 2 hours before which measurements cannot be made. CGM sensor will be applied on consented patients about 2.5 hours prior to surgery. The CGM monitor will be configured to not display the glucose measurements and trends (blinded mode). Lastly, the CGM clock will be synchronized to the hospital computer clock.

During surgery:

The institutional protocol for glucose management will be followed using the POC and lab glucose measurements as reference. The measurements made by the CGM will be blinded and the anesthesia provider will not be able to see or use the CGM values for clinical care. In the OR, the CGM monitor will placed on top platform of the anesthesia machine beside the POC glucose meter base. This location will ensure that the monitor is within 20 feet of the sensor and within the control of the anesthesia providers. Hourly blood glucose measurements performed by the POC glucose meter (Roche Diagnostics Inform II) or laboratory meter (part of arterial blood gas panel) will be automatically acquired and documented in the electronic anesthesia record. The CGM keeps a log of the continuous glucose measurements every 5 minutes for retrospective download and review. The anesthesia information system will also document the patient demographics (Age, Gender, BMI, etc), medications and fluid, anesthetic agent's concentrations, temperature, surgical and anesthesia events. These data elements can be retrospectively downloaded for analysis.

After surgery (PACU/ICU/Wards):

The institutional protocol for glucose management will be continued after surgery in PACU, surgical ICU or surgical wards. Glucose will continue to be monitored every 1-6 hours. In addition to POC measurements, blood samples taken for venous or arterial collection will be automatically documented in the inpatient electronic medical record. The CGM measurements will continue to be blinded to the nurse practitioner. CGM use will be continued for a total period of 72 hours after surgery or until the patient is discharged from the hospital whichever occurs earlier.

CGM monitor disconnect & cleaning:

The CGM sensor and monitor will be removed at the end of the study period by either the research coordinator or the bedside nurse. The CGM will be covered in a protective shield and cleaned per procedures approved for the CGM. After cleaning procedures are complete the monitor will be used on a new patient. Additionally, the CGM measurements will be downloaded by the principal investigator into a data file for later analysis.

Safety and feasibility check:

A safety and feasibility check will be performed after the CGM has been applied on 4 patients. The primary outcome measure at the safety check point will be the ability of the sensor to make measurements and transmit the results to the monitor without data drops (without significant interruptions during electrocautery and other surgical interventions, anesthetic interventions and medication administration). Additionally, the feasibility of applying, maintaining and using the sensor in an OR environment will be evaluated for any potential issues. Lastly, the study will also observe any unexpected incidence of patient safety issues - potential infection, rash, or swelling of the area where the sensor is applied, potential RF interference etc.

The study will be continued only after successful completion of the safety check, and only if there is reasonable assurance that the CGM can be used safely and reliably in the operating room and postoperative areas with acceptable accuracy (Mean Absolute Relative Difference ~ 20%) without significant interference from anesthetic drugs, electrocautery, edema and other surgery and anesthesia factors.

Data extraction and analysis:

The CGM glucose measurements made every 5 minutes will be downloaded from the monitor to a computer file using a software program provided by Dexcom Inc. Patient demographics (Age, Gender, BMI, DM status), preoperative labs (glucose, HbA1c), anesthesia and surgery events, POC glucose measurements, medication data (including insulin), temperature and anesthetic agent information will be extracted from the Anesthesia Information Management System (AIMS) database. Post-operative glucose measurements and medication information will be collected from Hospital Electronic Medical Record and Data warehouse system (AMALGA, Microsoft Inc. Redmond, WA).

Data analysis will focus on three aspects:

1. Test of equivalence:

   Paired CGM-POC measurements will be compared to determine mean bias (mean difference) and SD. The investigators will report the 95% limits of agreement, calculated as mean bias ± 1.96 X SD, the recommended statistic for assessing agreement between two methods of measurement. Data will be presented on Bland-Altman plots.
2. CGM accuracy and bias:

   The CGM measurements will be compared against the corresponding POC glucose measurements to evaluate accuracy. MARD (Mean Absolute Relative Difference) will be used as the main accuracy measure. Effect of confounding factors - body temperature, BMI, Diabetes status, inotrope score, anesthetic agents, medications and use of electrocautery on CGM functionality and measurement accuracy will be evaluated.

   CGM accuracy assessment will be performed via the following steps:
   * Pearson correlation coefficient between the CGM and POC glucose paired values
   * Clarke Error Grid analysis relating CGM-POC glucose measurement pairs to evaluate clinical accuracy (% measurements in zones A & B)
   * MARD ranges for all paired CGM-POC glucose measurements for the following glucose ranges <100, 100-140, 140-180, > 180 mg/dL
3. Trends and changes in blood glucose levels:

Trends and changes in blood glucose levels through the course of surgery and immediate postoperative phase (24 hours) will be analyzed across patients to determine consistent trend indicators (anesthesia and surgery events, use of medications, anesthetic agents etc). Specifically, multivariate analysis of glucose trends adjusted for covariates will be conducted to determine the effect of surgical stress, anesthesia and medications on blood glucose levels. CGM measurements will be used to evaluate the percentage of time glucose levels are within the desired range (100-140 mg/dL and 100-180 mg/dL) and evaluate the level of glucose excursions between hourly POC glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) diabetic (both Type 1 & 2) patients who are self-monitoring glucose levels (via finger stick measurements) two to three times daily.
* Scheduled to have elective general surgery at UW Medical Center. Preferably target Surgery A- Orthopedic/GYN surgery/Bariatric patients.
* Proposed case duration > 2 hour case.

Exclusion Criteria:

* Pregnant and lactating females
* MRI, CT & Diathermy procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irl B Hirsch, MD, Study Chair — University of Washington; David Flum, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CGM Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all participants at baseline are included in analysis
Arm/Group | CGM Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline A1C [Mean (Standard Deviation); unit: mmol/mol] | 57.4 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility Evaluation - Number of Unanticipated Safety Issues
Description: After CGM has been applied on the first 4 patients, the study team will evaluate the safety and feasibility of using CGM. Specifically, the team will check whether there are unanticipated adverse events such as rashes or discomfort
Time Frame: After 4 patients (2 months)
Population: Safety was assessed after 4 participants were enrolled; MARD was assessed after 10 participants were enrolled. The study stopped enrollment earlier than planned.
Measure: Number; unit: Number of unanticipated safety events
Arm/Group | CGM Patients
Number analyzed (Participants) | 4
Number of unanticipated safety events | 0

2. Primary Outcome: Mean Absolute Relative Difference for CGM and POC Glucose Measurements
Description: Compare glucose measurements made by a Dexcom G4 Professional Continuous Glucose Monitor (CGM) against point of care glucose meter (Accu-Check Inform II, Roche Diagnostics), during the intraoperative and postoperative phases. Measured as mean absolute relative difference (MARD) for CGM glucose values compared with the POC glucose measurements.
Time Frame: 10 months
Population: One patient was excluded from analysis due to incorrect insertion protocol.
Measure: Mean (Standard Deviation); unit: % of mean absolute relative difference
Arm/Group | CGM Patients
Number analyzed (Participants) | 9
% of mean absolute relative difference | 9.4 (7.7)

3. Primary Outcome: Feasibility of Instrument: Count of CGM Instrument Issues
Description: After 4 participants (2 months), the study team will assess the number of instrument breaks
Time Frame: After 4 participants (2 months)
Measure: Number; unit: number of instrument breaks
Arm/Group | CGM Patients
Number analyzed (Participants) | 4
number of instrument breaks | 0

ADVERSE EVENTS:
Time Frame: Surgery through up to 10 days after surgery or until the patient is discharged from the hospital whichever occurs earlier.
Arm/Group | CGM Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02572856/Prot_000.pdf